CLINICAL TRIAL: NCT00463203
Title: Bevacizumab and Irinotecan for Patients With Primary Brain Tumors and Progression After Standard Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Ulrik Lassen, Rigshospitalet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BI-Brain-01
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Brain Neoplasms; Glioma
Keywords: primary malignant brain tumor; grade II glioma; meningeoma; ependymoma; Recurrence or progression after standard treatment
MeSH Terms: conditions — Brain Neoplasms; Glioma; Ependymoma; Recurrence | interventions — Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg every 2 weeks
Drug: Irinotecan — 125 mg/m2 non-EIAED or 340 mg/m2 EIAED every 2 weeks

SUMMARY:
Irinotecan has demonstrated activity in malignant gliomas in multiple phase II studies. The activity is limited, with an approximately 15 % response rate and a progression-free survival of 3-5 months. Given the synergy between irinotecan and bevacizumab in colorectal cancer, and the high-level expression of vascular endothelial growth factor on malignant gliomas, one would expect synergy between bevacizumab and irinotecan against gliomas.

Recent data form a small study of 32 patients from Duke University have achieved a response rate of 62% in patients with malignant gliomas. Most included patients had glioblastomas, but this regimen may also have activity in more rare primary malignant brain tumors. The investigators therefore plan to include other primary malignant brain tumors in this study, and the clinical activity will be correlated with biomarkers and PET results of metabolic activity and blood flow. This may result in information that can be used to individualize therapy in the future.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Histological verification of primary malignant brain tumor, or grade II glioma, meningeoma or ependymoma with progression and no other treatment options (including brain stem gliomas without histological verification)
* Recurrence or progression after standard treatment (debulking surgery of possible, radiotherapy and for grade III or IV tumors temozolomide or other chemotherapy.
* Evidence of measurable recurrent progressive disease (CT/MRI scan)
* An interval of at least 4 weeks between prior surgical resection and study enrollment
* An interval of at least 4 weeks between prior radiotherapy or chemotherapy and enrollment on this protocol.
* PS 0-2 (ECOG scale)
* Age > 18
* Life expectancy > 3 month
* Normal organ function:
* Platelets > 125 x 109/l
* Hemoglobin >6,2 mmol/l
* Leukocytes > 3 x 109/l
* ACN> 1,5 x 109/l
* ASAT or ALAT < 3 x upper normal limit
* Bilirubin < 1,5 x upper normal limit
* Creatinine clearance > 45 ml/min
* APTT < normal limit
* INR < normal limit
* Fertile females must use oral contraceptive, IUD (intrauterine device), gestagen sustained release injection, subdermal implantation, transdermal patch or hormonal vaginal ring. This must continue at least three months after the patients is off-study. Fertile males must use preservatives
* No sign of cerebral bleeding

Exclusion criteria:

* Radiotherapy or chemotherapy within the last 4 weeks.
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Prior VEGF-based therapy
* Any condition (medical, social, psychological), which would prevent adequate information and follow-up
* Any other concurrent active malignancy, except, adequately treated basal or squamous cell carcinoma of the skin, or carcinoma in situ.
* Any significant cardiac disease (New York Heart Association Class II or greater), arrhythmia, congestive heart failure, acute myocardial infarction within 6 months or unstable angina pectoris.
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis, coagulopathy or taking ASA, NSAIDs or clopidogrel
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0, anticipation of need for major surgical procedure during the curse of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 0
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 month prior to day 0
* History of known HIV, Hepatitis B and Hepatitis C negative
* Any ongoing infection, uncontrolled diabetes mellitus, serious non-healing wound, ulcer or bone fracture
* Pregnancy or breast feeding
* Requires therapeutic anti-coagulation
* Blood pressure > 150/100 mmHG
* Grade 2 or greater proteinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 6 months

SECONDARY OUTCOMES:
Response rate - Response according to MacDonald criteria | 6 months
Adverse event according to CTCAE 3.0 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD., PH.D., Principal Investigator — Rigshospitalet, Dept. of Oncology
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense